CLINICAL TRIAL: NCT07076238
Title: A Single-Center Observational Biomarker Investigation of Response to Bacteriophage Treatment for Bacterial Infection
Brief Title: Biomarkers of Phage Treatment Response in NTM and Other Infections
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 25-00062
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Nontuberculous Mycobacterial Lung Disease
Keywords: Bacteriophage therapy; Refractory bacterial infection
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, sputum samples, and oral rinse samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants receiving phage therapy: Participants who have a positive match for their Nontuberculous Mycobacterial (NTM) isolate will start on mycobacteriophage treatment. Blood and leftover and/or discarded airway samples will be obtained from follow up visits of patients.
  Interventions: Biological: Bacteriophage Treatment
- Participants not receiving phage therapy: Participants who don't have a positive match and/or do not start on mycobacteriophage treatment. Blood and leftover and/or discarded airway samples will be obtained from follow up visits of patients.

INTERVENTIONS:
Biological: Bacteriophage Treatment — Participants who have a positive match for their NTM isolate will start on mycobacteriophage treatment per prescribed treatment regimen.
  Groups: Participants receiving phage therapy

SUMMARY:
This study aims to identify biomarkers associated with response to phage therapy for refractory bacterial infections. This includes mycobacteriophage treatment for patients with nontuberculous mycobacterial infections. Blood and airway samples will be obtained from follow up visits of patients with refractory bacterial infections that are considered for phage therapy. Samples will be compared between those that receive phage therapy and those that did not. Biomarkers will include changes in the airway microbiome, transcriptome, inflammatory cytokines, and development of neutralizing antibody against phages. The primary endpoint is to identify biomarkers associated with clinical and/or radiographic improvement and/or culture improvement which includes clearing of cultures or decrease in qualitative or resolution of signs and symptoms of infection after at least 6-8 weeks of bacteriophage therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older
2. Provision of appropriate written consent
3. Willingness and ability to participate in study procedures
4. Diagnosis of bacterial/mycobacterial infection that meets criteria for treatment (clinical, radiographic, and microbiologic data)
5. Patients are being considered by clinician for phage therapy as a part of their standard of care

Exclusion Criteria:

1. Patients under 18 years of age
2. Pregnant individuals as this population is not considered for phage treatment due to unknown risks of the treatment
3. Breastfeeding Individuals who are breastfeeding as this population is not considered for phage treatment due to unknown risk to the infant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Nontuberculous Mycobacterial (NTM) disease who are considered for treatment with phage therapy will be recruited. Those that have a positive match for their NTM isolate and starts on mycobacteriophage treatment will be considered cases while those that do not have a positive match and/or does not start on mycobacteriophage treatment will be considered controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2030-06-25 (Estimated); Study Completion 2032-06-25 (Estimated)

PRIMARY OUTCOMES:
Biomarkers associated with clinical and/or radiographic improvement and/or culture improvement | End of study (up to 2 years)
  Improvement includes clearing of cultures or decrease in qualitative or resolution of signs and symptoms of infection after at least 6-8 weeks of bacteriophage therapy.

SECONDARY OUTCOMES:
Biomarkers associated with the development of neutralization antibodies | End of study (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Addrizzo-Harris, MD, FCCP, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 3 months and ending 5 years following article publication, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Doreen.Addrizzo@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Doreen.Addrizzo@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.